CLINICAL TRIAL: NCT06594224
Title: Comparison of IV Nalbuphine Versus Ibuprofen for Postoperative Pain Control in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, RESnTEC, Institute of Research, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NishterMultan-1
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Ibuprofen; Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Ibuprofen Group (Experimental): Females in this group (n=40) were given 800 mg Ibuprofen in 200 cc normal saline intravenously at the time of arrival in the ward
  Interventions: Drug: Ibuprofen
- IV Nalbuphine (Experimental): Patients in this group received 20 mg nalbuphine in 200 cc normal saline IV at the time of arrival in the ward.
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Ibuprofen — Patients were given 800 mg Ibuprofen in 200 cc normal saline intravenously at the time of arrival in the ward.
  Arms: IV Ibuprofen Group
Drug: Nalbuphine — Patients received 20 mg nalbuphine in 200 cc normal saline IV at the time of arrival in the ward.
  Arms: IV Nalbuphine

SUMMARY:
The local data is insufficient to directly compare IV nalbuphine versus ibuprofen among people in this region. The findings of this study would add to the existing data and would be helpful for health providers to opt for a better option for postoperative pain relief following a cesarean section under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Parturient females
* Aged between 18-45 years
* Gestational age above 32 weeks
* ASA class I to II
* Anticipated hospital stay for at least 24 hours

Exclusion Criteria:

* Known allergy to the drugs being evaluated in this study
* Renal and/or hepatic impairment (as per medical record)
* History of bronchial asthma or history or risk of intracranial hemorrhage (as per medical record)
* Low platelets count (<70000) or with bleeding diathesis
* BMI above 30 kg/m2

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy in pain control | At 1 hour, 3 hours, and 6 hours.
  Outcome was noted in the form of VAS pain scores. Scores from 1 to 3 were labeled as mild pain, 4 to 6 as moderate pain, and 7 to 10 as severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mehnaz Khakwani, FCPS, Principal Investigator — Department of Obstetric and Gynecology Nishtar Medical University, Multan; Hajra Sultana, FCPS, Principal Investigator — Department of Obstetric and Gynecology Nishtar Medical University, Multan
Locations (2):
- Pakistan (2):
  - Nishtar Hospital, Multan, Punjab Province
  - Nishtar Medical University, Multan, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request

REFERENCES:
- [Derived] Khakwani M, Parveen R, Sultana H. Comparison of IV Nalbuphine versus ibuprofen for Postoperative Pain control in cesarean section. Pak J Med Sci. 2025 Sep;41(9):2612-2617. doi: 10.12669/pjms.41.9.11016. PMID 41070313